## **LEAD IT!**

## An App to Enable Persons With Early Stage Dementia to Lead Group Activities for Their Peers

Project Also Known As:

PEER: Purposeful Engagement for Every Resident

NCT05516342

Statistical Analysis Plan

Last Updated: 8/3/2023

The statistical design used for this project will be tied to the one relevant Specific Aim: Examine the effects of resident-led LEAD IT! on people with dementia. The Cluster Randomized Trial (CRT) that will be implemented during this project entails the use of a two-way mixed design ANOVA, with a between-subjects factor of Group (CG vs. TG) and within-subjects factor of Time (baseline versus treatment (proximal measures) or posttreatment (distal measures)). To examine engagement, multiple observations of participants will be taken at both baseline and treatment using the Menorah Park Engagement Scale (MPES). Then, means will be calculated for each participant for each item (type of engagement / affect) on the MPES. For MPES data, we anticipate detecting a Group x Time interaction effect, with TG participants exhibiting significantly greater increases in constructive engagement and pleasure at treatment, as compared to CG participants. For distal measures, we anticipate detecting a Group x Time interaction effect, with TG participants exhibiting significantly greater increases in DEMQOL scores at treatment, as compared to CG participants. We anticipate TG participants will exhibit significantly greater decreases in GDS-SF, CMAI, and/or NPI-NH scores at treatment, as compared to CG participants.